CLINICAL TRIAL: NCT01592916
Title: Acute Effects of Exercise in Women With FM
Brief Title: Acute Effects of Exercise in Women With Fibromyalgia (FM)
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: GU-143-12
Record Dates: First submitted 2012-05-04; First posted 2012-05-07 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain; Women; Exercise; IGF1
MeSH Terms: conditions — Fibromyalgia; Pain; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fibromyalgia: Women with fibromyalgia, aged 20-50 years
- Healthy controls: Women without severe disease, aged 20-50 years

SUMMARY:
The investigators previous studies of aerobic exercise in women with fibromyalgia (FM) have shown that exercise improves body functions and/or symptom severity in most patients, but not in all. About a third of patients with FM have been shown to have low levels of IGF-1. The purpose of this project is to study individual and biological factors that interact with outcomes of short-term (acute) exercise in FM.

Method. A controlled prospective exercise study. Thirty women with FM and 30 healthy age-matched women, aged 20-50 years, will be recruited to the study. Two 15-minute ergometer bicycle exercise tests will be conducted in feasting patients, separated by one month. The first exercise test is at a low and the second at a high intensity. Measurements comprise blood test, pain rating and pain threshold, conducted before and after the test. The levels of IGF-1, IL-6 and IL-8 will be measured, and the changes in them will be related to health status and pain.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of fibromyalgia
* age 20-50 years

Exclusion Criteria:

* heart disease
* neurological disease
* severe osteoarthritis

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants are recruited from previous studies.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-05-10 (Actual); Primary Completion 2012-11-23 (Actual); Study Completion 2012-11-23 (Actual)

PRIMARY OUTCOMES:
IGF1 level | 15 min
  Ergometer cycle test of 15 minutes at low respective high intensity. Blood test is done before and after exercise. Change in quantity of IGF1 is measured.

SECONDARY OUTCOMES:
Pain rating | 15 minutes
  Pain is rated by the test person before and after the ergometer cycle test.
Pain threshold | 15 minutes
  Pain threshold is measured before and after the ergometer test.
Interleukin 6 and 8 | 15 minutes
  Blood test is done before and after the ergometer bicycle test. Quantity of interleukin 6 and 8 is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Mannerkorpi, Assoc prof, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Dept of Physical Therapy, Gothenburg, Sweden

REFERENCES:
- [Result] Mannerkorpi K, Landin-Wilhelmsen K, Larsson A, Cider A, Arodell O, Bjersing JL. Acute effects of physical exercise on the serum insulin-like growth factor system in women with fibromyalgia. BMC Musculoskelet Disord. 2017 Jan 25;18(1):37. doi: 10.1186/s12891-017-1402-y. PMID 28122522